CLINICAL TRIAL: NCT02207088
Title: An Open-Label Study to Evaluate the Safety and Efficacy of Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir With or Without Ribavirin (RBV) in Adults With Genotype 1 Chronic Hepatitis C Virus (HCV) Infection, With Severe Renal Impairment or End-Stage Renal Disease (RUBY-I)
Brief Title: Ombitasvir/ABT-450/Ritonavir and Dasabuvir With or Without Ribavirin in HCV Genotype 1-Infected Adults With Chronic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-226; 2014-001527-77 (EudraCT Number)
Record Dates: First submitted 2014-07-31; First posted 2014-08-01 (Estimated); Results first posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-10

CONDITIONS: Chronic Hepatitis C; Hepatitis C Virus; Compensated Cirrhosis; Severe Renal Impairment; End-stage Renal Disease
Keywords: Chronic Hepatitis C; Hepatitis C; End-stage renal disease; Hepatitis C Genotype 1; Severe Renal Impairment; renal disease; Compensated Cirrhosis; Renal impairment; dialysis; Hepatitis C Virus; cirrhosis
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Renal Insufficiency; Kidney Failure, Chronic; Kidney Diseases; Fibrosis | interventions — ombitasvir; Viekira Pak; paritaprevir; dasabuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 3-DAA (Direct Acting Antivirals) with or without RBV (Experimental): 3-DAA (ombitasvir/paritaprevir/ritonavir 25 mg/150 mg/100 mg once daily [QD] and dasabuvir 250 mg twice daily [BID]) with or without ribavirin (RBV; dosed divided twice a day) for 12 or 24 weeks
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir; Drug: dasabuvir; Drug: Ribavirin

INTERVENTIONS:
Drug: ombitasvir/paritaprevir/ritonavir — tablet
  Other Names: ABT-450/r/ABT-267; Viekira Pak; paritaprevir also known as ABT-450; ombitasvir also known as ABT-267; dasabuvir also known as ABT-333
Drug: dasabuvir — tablet
  Other Names: ABT-333
Drug: Ribavirin — tablet
  Other Names: RBV

SUMMARY:
This open-label study will evaluate safety, pharmacokinetics and efficacy of a 12 or 24-week regimen of ombitasvir/paritaprevir/ritonavir and dasabuvir with or without ribavirin in HCV-genotype 1-infected subjects with an Estimated Glomerular Filtration Rate (eGFR) <30, including those on hemodialysis or peritoneal dialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Positive for anti-HCV Ab (Antibody) and HCV RNA >1,000 IU/mL at Screening.
2. Screening laboratory result indicating HCV genotype 1 infection.
3. Subject has never received antiviral treatment for hepatitis C infection (treatment-naive subject) or subject has received previous treatment with peginterferon with or without RBV with non-response (HCV RNA quantifiable at end of treatment or relapsed after end of treatment).
4. Estimated Glomerular Filtration Rate (eGFR) < 30 mL/min/1.73 m^2 as estimated by the Modification of Diet in Renal Disease (MDRD) method.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding.
2. Positive test result for Hepatitis B surface antigen (HBsAg) or anti-Human Immunodeficiency Virus (HIV Ab).
3. Any current or past clinical evidence of Child-Pugh B or C classification or clinical history of liver decompensation such as ascites (noted on physical exam), variceal bleeding, or hepatic encephalopathy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-09-23 (Actual); Primary Completion 2016-12-06 (Actual); Study Completion 2016-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Cohen, MD, Study Director — AbbVie

REFERENCES:
- [Derived] Shuster DL, Menon RM, Ding B, Khatri A, Li H, Cohen E, Jewett M, Cohen DE, Zha J. Effects of chronic kidney disease stage 4, end-stage renal disease, or dialysis on the plasma concentrations of ombitasvir, paritaprevir, ritonavir, and dasabuvir in patients with chronic HCV infection: pharmacokinetic analysis of the phase 3 RUBY-I and RUBY-II trials. Eur J Clin Pharmacol. 2019 Feb;75(2):207-216. doi: 10.1007/s00228-018-2566-6. Epub 2018 Oct 5. PMID 30291369
- [Derived] Pockros PJ, Reddy KR, Mantry PS, Cohen E, Bennett M, Sulkowski MS, Bernstein DE, Cohen DE, Shulman NS, Wang D, Khatri A, Abunimeh M, Podsadecki T, Lawitz E. Efficacy of Direct-Acting Antiviral Combination for Patients With Hepatitis C Virus Genotype 1 Infection and Severe Renal Impairment or End-Stage Renal Disease. Gastroenterology. 2016 Jun;150(7):1590-1598. doi: 10.1053/j.gastro.2016.02.078. Epub 2016 Mar 11. PMID 26976799

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The intent-to-treat (ITT) population consisted of all enrolled participants who received at least 1 dose of study drug.
Groups:
- 3-DAA ± RBV: 3-DAA (ombitasvir/paritaprevir/ritonavir 25 mg/150 mg/100 mg once daily [QD] and dasabuvir 250 mg twice daily [BID]) with or without ribavirin (RBV; dosed divided twice a day) for 12 or 24 weeks
Period: Overall Study
Arm/Group | 3-DAA ± RBV
Started | 68
Completed | 66
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: Safety and demographic analyses were performed on safety population, which is the same as the ITT population.
Groups:
- 3-DAA ± RBV: 3-DAA (ombitasvir/paritaprevir/ritonavir 25 mg/150 mg/100 mg once daily [QD] and dasabuvir 250 mg twice daily [BID]) with or ribavirin (RBV; dosed divided twice a day) for 12 or 24 weeks
Arm/Group | 3-DAA ± RBV
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (7.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 57

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 (SVR12) Weeks Post-treatment
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification (<LLOQ) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last actual dose of study drug
Population: All randomized participants who received at least one dose of study drug (ITT population).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3-DAA ± RBV
Number analyzed (Participants) | 68
percentage of participants | 94.1 [85.8 to 97.7]

2. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as confirmed HCV RNA ≥ LLOQ after < LLOQ during treatment, confirmed increase of > 1 log (subscript)10(subscript) IU/mL above the lowest value post-baseline HCV RNA during treatment, or HCV RNA ≥ LLOQ persistently during treatment with at least 6 weeks of treatment.
Time Frame: Up to 24 weeks
Population: All randomized participants who received at least one dose of study drug (ITT population).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3-DAA ± RBV
Number analyzed (Participants) | 68
percentage of participants | 0 [0.0 to 5.3]

3. Secondary Outcome: Percentage of Participants With Post-Treatment Relapse
Description: Post-treatment relapse was defined as confirmed HCV RNA ≥ LLOQ between end of treatment and 12 weeks after the last dose of study drug among participants completing treatment and with HCV RNA < LLOQ at the end of treatment.
Time Frame: Within 12 weeks after the last dose of study drug
Population: All randomized participants who received at least one dose of study drug (ITT population) with HCV RNA < LLOQ at the end of treatment and completed treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 3-DAA ± RBV
Number analyzed (Participants) | 65
percentage of participants | 1.5 [0.3 to 8.2]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the time of study drug administration until 30 days after the last dose of study drug (up to 28 weeks).
Description: TEAEs and TESAEs are defined as any adverse event (AE) with an onset date that is after the first dose of study drug until 30 days after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Groups:
- 3-DAA +/- RBV: 3-DAA (ombitasvir/paritaprevir/ritonavir 25 mg/150 mg/100 mg once daily [QD] and dasabuvir 250 mg twice daily [BID]) with or without ribavirin (RBV; dosed divided twice a day) for 12 or 24 weeks
Arm/Group | 3-DAA +/- RBV
Serious Adverse Events (participants affected / at risk) | 17/68
Other Adverse Events (participants affected / at risk) | 51/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3-DAA +/- RBV (N=68)
ANAEMIA (Blood and lymphatic system disorders) | 1
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1
ANGINA PECTORIS (Cardiac disorders) | 1
CARDIAC ARREST (Cardiac disorders) | 1
CARDIAC TAMPONADE (Cardiac disorders) | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 1
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 1
DYSPHAGIA (Gastrointestinal disorders) | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1
VOLVULUS (Gastrointestinal disorders) | 1
LIVER INJURY (Hepatobiliary disorders) | 1
ARTERIOVENOUS GRAFT SITE INFECTION (Infections and infestations) | 1
INTERVERTEBRAL DISCITIS (Infections and infestations) | 1
PERITONITIS BACTERIAL (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 2
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1
SYNCOPE (Nervous system disorders) | 1
MENTAL STATUS CHANGES (Psychiatric disorders) | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
ACCELERATED HYPERTENSION (Vascular disorders) | 1
HYPERTENSIVE CRISIS (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3-DAA +/- RBV (N=68)
ANAEMIA (Blood and lymphatic system disorders) | 26
DIARRHOEA (Gastrointestinal disorders) | 13
NAUSEA (Gastrointestinal disorders) | 13
VOMITING (Gastrointestinal disorders) | 10
FATIGUE (General disorders) | 20
OEDEMA PERIPHERAL (General disorders) | 5
HAEMOGLOBIN DECREASED (Investigations) | 9
DECREASED APPETITE (Metabolism and nutrition disorders) | 6
DIZZINESS (Nervous system disorders) | 6
HEADACHE (Nervous system disorders) | 8
PRURITUS (Skin and subcutaneous tissue disorders) | 8
HYPERTENSION (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.